CLINICAL TRIAL: NCT03887078
Title: Randomized Trial of an Innovative Smartphone Application for Bariatric Surgery
Brief Title: Noom Coach for Bariatric Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noom Inc. (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R44DK116370 (NIH)
Record Dates: First submitted 2019-03-17; First posted 2019-03-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Obesity; Bariatric Surgery; mHealth
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Two successive randomizations based on patterned response to primary intervention. Pre-surgical participants (n=200) will be randomized to groups in Noom Coach for Bariatric Health or standard care pre-surgery. Post-surgery, optimal and suboptimal responders will be randomized to Noom Bariatric or standard care. This design allows for comparisons between all 8 conditions. Contrasts allow us to answer the critical question about main effects of Noom Pre-surgery and Noom augmentation and whether this augmentation effect differs based on empirically derived classification of early response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- A. Presurgery Noom Bariatric + Augmentation Noom Bariatric (Experimental): Self-monitoring will be conducted through Noom Coach for Bariatric Health, and individuals will receive a specialized set of instructions on how to use the app. Intervention responsive individuals will be randomized post-surgery to Noom Bariatric augmentation.
  Interventions: Behavioral: Noom Coach for Bariatric Health
- B. Presurgery Noom Bariatric + Augmentation Standard Care (Experimental): Self-monitoring will be conducted through Noom Coach for Bariatric Health, and individuals will receive a specialized set of instructions on how to use the app. Intervention responsive individuals will be randomized post-surgery to "usual care" in which participants are free to seek any assistance for their bariatric post-surgery care during the study period.
  Interventions: Behavioral: Noom Coach for Bariatric Health
- C. Presurgery Noom Bariatric + Augmentation Noom Bariatric (Experimental): Self-monitoring will be conducted through Noom Coach for Bariatric Health, and individuals will receive a specialized set of instructions on how to use the app. Intervention non-responsive individuals will be randomized post-surgery to Noom Bariatric augmentation.
  Interventions: Behavioral: Noom Coach for Bariatric Health
- D. Presurgery Noom Bariatric + Augmentation Standard Care (Experimental): Self-monitoring will be conducted through Noom Coach for Bariatric Health, and individuals will receive a specialized set of instructions on how to use the app. Intervention non-responsive individuals will be randomized post-surgery to "usual care" in which participants are free to seek any assistance for their bariatric post-surgery care during the study period.
  Interventions: Behavioral: Noom Coach for Bariatric Health
- E. Pre-surgery Standard Care + Augmentation Noom Bariatric (Experimental): The control group will be a "usual care" condition in which participants are free to seek any assistance for their bariatric surgery care during the study period. Usual care responsive individuals will be randomized post-surgery to Noom Bariatric augmentation.
  Interventions: Behavioral: Noom Coach for Bariatric Health
- F. Pre-surgery Standard Care + Augmentation Standard Care (No Intervention): The control group will be a "usual care" condition in which participants are free to seek any assistance for their bariatric surgery care during the study period. Usual care responsive individuals will be randomized post-surgery to usual care.
- G. Pre-surgery Standard Care + Augmentation Noom Bariatric (Experimental): The control group will be a "usual care" condition in which participants are free to seek any assistance for their bariatric surgery care during the study period. Usual care non-responsive individuals will be randomized post-surgery to Noom Bariatric augmentation.
  Interventions: Behavioral: Noom Coach for Bariatric Health
- H. Pre-surgery Standard Care + Augmentation Standard Care (No Intervention): The control group will be a "usual care" condition in which participants are free to seek any assistance for their bariatric surgery care during the study period. Usual care non-responsive individuals will be randomized post-surgery to usual care.

INTERVENTIONS:
Behavioral: Noom Coach for Bariatric Health — Noom Coach for Bariatric Health offers a sustainable, low-cost, coach-led intervention, and an innovative solution to issues with pre-bariatric surgery weight loss. The intervention will take place over 8 weeks pre and or post-surgery.
  Arms: A. Presurgery Noom Bariatric + Augmentation Noom Bariatric; B. Presurgery Noom Bariatric + Augmentation Standard Care; C. Presurgery Noom Bariatric + Augmentation Noom Bariatric; D. Presurgery Noom Bariatric + Augmentation Standard Care; E. Pre-surgery Standard Care + Augmentation Noom Bariatric; G. Pre-surgery Standard Care + Augmentation Noom Bariatric

SUMMARY:
Mobile technologies/smartphone applications offer a means to effect behavior change without significant obstacles that typically limit implementation of empirically supported therapies (e.g., in-person sessions); however, rigorous research on apps is limited, and high-quality, adequately powered, randomized controlled trials with large samples are required. As more Americans consider bariatric surgery for the treatment of severe obesity, it is imperative to improve factors influencing suboptimal surgical outcomes (e.g., failure to adhere to diet and exercise recommendations and psychosocial impairment). This study will evaluate the effect of the Noom Coach for Bariatric Health platform in improving standard interventions utilized in bariatric surgery programs.

DETAILED DESCRIPTION:
Overweight and obesity have reached epidemic proportions in the United States. As few behavioral treatments are effective for weight loss, bariatric surgery is an increasingly important option. Although these procedures are more helpful than psychosocial treatments, post-operative weight losses vary widely, and a notable subset of patients demonstrate suboptimal weight loss or substantial weight regain. Adherence to treatment recommendations is a likely contributor to these variable outcomes. Smartphone applications (apps) designed to augment behavior change or enhance adherence, have expanded exponentially in recent years, and are a potentially useful option to improve outcomes, but rigorous research on apps is limited, and high-quality, adequately powered, randomized controlled trials with large samples are required. This study will test a combined smartphone app and health coaching system to improve adherence and behavioral/psychosocial outcomes for patients receiving bariatric surgery. The aims have not been modified since the original phase 1 and will compare usual pre-operative care and pre-surgical use of Noom Coach for Bariatric Health on post-surgery adherence and psychosocial variables in a larger test (n=200) to explore whether usage of the app is a viable predictor of subsequent post-operative weight trajectories 12 months following surgery. This study will also examine app usage as a viable predictor of subsequent post-operative weight and psychosocial trajectories in the 12 months post-surgery and establish sensitivity and specificity of early optimal response to surgical intervention using weight loss, diet and exercise adherence, and psychosocial adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in: (1) the Metabolic, Endocrine, and Minimally Invasive Surgery Division at Mount Sinai and planning to receive a bariatric procedure.
* Between the ages of 18 and 60 at entry to the study.
* Speak English.

Exclusion Criteria:

* Clinically significant cognitive limitations (Wechsler Abbreviated Scale of Intelligence IQ Estimate < 70) or history of developmental disability.
* History of neurological disorder or injury (e.g., seizure disorder or moderate or severe head injury with >10 minutes loss of consciousness).
* Current/lifetime DSM-5 bipolar disorder, schizophrenia, or psychotic disorder.
* Acute suicide risk.
* Current DSM-5 alcohol or substance use disorder.
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Change in adherence to dietary recommendations | Baseline, 8 weeks, 3 months, and 12 months
  Change in adherence to recommendations provided within pre-bariatric surgery program will be assessed using the ASA-24 interview. The interview is a 24-hr recall of all food and drink consumed. This interview will serve as the basis for measuring the adherence to dietary recommendations.
Change in adherence to physical activity recommendations (Activity Tracker) | Baseline, 8 weeks, 3 months, and 12 months
  Change in adherence to physical activity recommendations will be measured using information collected from each participants activity tracker (FitBit). The activity tracker records number of steps taken each day and any physical activity performed.
Change in adherence to physical activity recommendations (IPAQ) | Baseline, 8 weeks, 3, 6, 9, and 12 months
  Change in adherence to physical activity recommendations will also be measured using self reported physical activity using the International Physical Activity Questionnaire (IPAQ) The IPAQ is a 27- item questionnaire that assesses physical activity over the past week as a part of everyday activity, activity as a part of work, and activity as recreation. Scores include both minutes and days spent doing physical activity with higher scores indicating more time spent doing these activities. The measure can be scored categorically (low, moderate, high) or continuously using a defined scoring protocol.
Anthropometric changes (weight) | Baseline, 8 weeks, 3, 6, and 12 months
  To calculate trajectories of BMI, measures of height (inches) and weight (pounds) will be obtained at all in-person visits.
Anthropometric changes (height) | Baseline, 8 weeks, 3, 6, and 12 months
  To calculate trajectories of BMI, measures of height (inches) and weight (pounds) will be obtained at all in-person visits.

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline, 8 weeks, 3, 6, 9, and 12 months
  Change in EDE-Q as compared to baseline. Questionnaire to assess for eating disorder symptomology. A 28 item measure with 4 subscales of restraint, eating concern, shape concern, and weight concern. Scores range from 0-168 with higher scores indicating more severe eating disorder pathology. Average scores on each subscale are used in addition to an average global score.
Depression Anxiety Stress Scales (DASS) | Baseline, 8 weeks, 3, 6, 9, and 12 months
  Change in symptoms of depression, anxiety, and stress from baseline. A 42-item self-report questionnaire assessing three related negative emotional states: depression, anxiety, and stress. Items are scored on a 0-3 Likert scale with ranges within each emotional state for normal, mild, moderate, severe and extremely severe symptoms. Higher scores indicate more severe symptoms. Ranges in severity are reported as sum scores for each emotion state. Depression includes normal (0-9), mild (10-13), moderate (14-20), severe (21-27), extremely severe (28+). Anxiety includes normal (0-7), mild (8-9), moderate (10-14), severe (15-19) extremely severe (20+) Stress includes normal (0-14), mild (15-18) , moderate (19-25), severe (26-33) extremely severe (34+).
Short Form-36 Health Survey (SF-36) | Baseline, 8 weeks, 3, 6, 9, and 12 months
  The SF-36 is a 10-item self-report of health-related quality of life measure that generates eight scaled scored. Individual items are scored 0-100 with higher scores indicating a more favorable health state. The eight subscales, reported as weighted means as (0-100) for each scale, include physical functioning, bodily pain, role limitations due to physical health, role limitations due to personal and emotional problems, emotional well being, social functioning, energy/fatigue, general health perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hildebrandt, PsyD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Andreas Michaelides, PhD, Principal Investigator — Noom Inc.
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No